CLINICAL TRIAL: NCT01960049
Title: Multicentre Evaluation of a Novel Technique of Analgesia Following Open Liver Resection: Medial Open Transversus Abdominis Plane (MOTAP) Catheters
Brief Title: Novel Technique of Analgesia Following Open Liver Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-0493-A
Record Dates: First submitted 2013-09-23; First posted 2013-10-10 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2016-05

CONDITIONS: Postoperative Pain; Liver Resection
Keywords: Postoperative pain; Liver resection; Medial Open Transversus Abdominis Plane catheter
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Analgesia, Patient-Controlled; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOTAP Catheter with Saline and IV PCA (Placebo Comparator): Control group will have saline 20cc of 0.9% normal saline injected into the catheters and then run at 5ml/hr for 72 hours
  Interventions: Procedure: saline and IV PCA
- MOTAP catheter with ropivocaine and IV PCA (Active Comparator): 20cc of 0.2% ropivacaine will be injected in two equal divided doses through the two catheters then run at 5ml/hr for 72 hours
  Interventions: Procedure: ropivacaine + iv PCA

INTERVENTIONS:
Procedure: ropivacaine + iv PCA
  Arms: MOTAP catheter with ropivocaine and IV PCA
Procedure: saline and IV PCA
  Arms: MOTAP Catheter with Saline and IV PCA

SUMMARY:
Abdominal wall incisions used for liver surgeries are associated with significant postoperative pain and disability. Epidural analgesia is often contraindicated in these patients due to common bleeding problems. Furthermore, drugs such as acetaminophen and opioids are often inadequate and can lead to detrimental side-effects. Abdominal wall (AW) catheters can be placed during surgical closure along the incision line and can be used to administer local anesthetics for postoperative pain. The study is a multi-centre, double-blind, randomized controlled trial involving 120 patients undergoing elective liver surgery. Patients will be randomly assigned to AW catheter group treated with drug or control treated with saline. Treatment group will receive AW catheters with ropivacaine plus standard patient controlled analgesia (PCA). Control group will obtain AW with normal saline and no local anesthetics and PCA. Patients are followed for 6 months post-operatively for pain scores, side-effects, chronic pain and complications.

ELIGIBILITY:
Inclusion Criteria:

* >18 years age
* Undergoing liver resection using a subcostal incision

Exclusion Criteria:

* Patients unable to comprehend instructions, consent, or co-operate with pain assessment (including psychiatric disorders, pre-operative sedation, coma)
* Allergy to any study medications
* Patient not able to be extubated postoperatively for any clinical reason
* Laparoscopic surgery
* Co-existing epidural or intrathecal analgesia
* Chronic pain disorders or on long-term opioid use
* History of substance or alcohol abuse
* Transplant donor liver resections
* Patients with liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | PCA opioid consumption every 12 hours for 72 hours as well as total opioid consumption for the entire hospital stay.
  The primary endpoint is mean cumulative postoperative opioid consumption over the first two postoperative days (48 hours). Both intravenous PCA opioids and oral opioids will be recorded from the patient's medical records daily, converted to morphine equivalents, and compared between the two groups.
  The following information will be collected at regular intervals as a measure of the primary endpoints: Cumulative i.v. PCA opioid consumption every 12 hours for 72 hours as well as total opioid consumption for the entire hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Hance Clarke, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario

REFERENCES:
- [Derived] Page MG, Karanicolas PJ, Cleary S, Wei AC, McHardy P, Ladak SSJ, Ayach N, Sawyer J, McCluskey SA, Srinivas C, Katz J, Coburn N, Hallet J, Law C, Greig P, Clarke H. In-hospital opioid consumption, but not pain intensity scores, predicts 6-month levels of pain catastrophizing following hepatic resection: A trajectory analysis. Eur J Pain. 2019 Mar;23(3):503-514. doi: 10.1002/ejp.1324. Epub 2018 Nov 8. PMID 30298685
- [Derived] Karanicolas PJ, Cleary S, McHardy P, Kiss A, Sawyer J, Behman R, Ladak S, McCluskey SA, Srinivas C, Katz J, Coburn N, Law C, Wei AC, Greig P, Hallet J, Clarke H. Medial Open Transversus Abdominis Plane (MOTAP) Catheters Reduce Opioid Requirements and Improve Pain Control Following Open Liver Resection: A Multicenter, Blinded, Randomized Controlled Trial. Ann Surg. 2018 Aug;268(2):233-240. doi: 10.1097/SLA.0000000000002657. PMID 29300708
- [Derived] Karanicolas P, Cleary S, McHardy P, McCluskey S, Sawyer J, Ladak S, Law C, Wei A, Coburn N, Ko R, Katz J, Kiss A, Khan J, Coimbatore S, Lam-McCulloch J, Clarke H. Medial open transversus abdominis plane (MOTAP) catheters for analgesia following open liver resection: study protocol for a randomized controlled trial. Trials. 2014 Jun 21;15:241. doi: 10.1186/1745-6215-15-241. PMID 24950773